CLINICAL TRIAL: NCT03506841
Title: Efficacy and Safety of Cerebrolysin on Neurodevelopmental Outcome of Preterm Infants
Brief Title: Cerebrolysin and Neurodevelopment in Preterm Infants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mansoura University Children Hospital (Other)
Responsible Party: Principal Investigator, Nehad Nasef, Professor of Pediatrics, Mansoura University Children Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Mansoura NICU 2016
Record Dates: First submitted 2018-04-13; First posted 2018-04-24 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Infant Development; Cerebral Palsy; Preterm Infant
MeSH Terms: conditions — Cerebral Palsy; Premature Birth | interventions — cerebrolysin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cerbrolysin (Active Comparator): Preterm infants with gestational age less than 32 weeks at birth will receive once weekly Cerebrolysin injections of 0.1 mL/kg body weight for 3 months (total of twelve injections) starting at the corrected postnatal age of 5 months.
  Interventions: Drug: Cerebrolysin
- Control (No Intervention): Preterm infants with gestational age less than 32 weeks at birth will receive routine care.

INTERVENTIONS:
Drug: Cerebrolysin — Cerebrolysin injections of 0.1 mL/kg body weight for 3 months (total of twelve injections).
  Arms: Cerbrolysin

SUMMARY:
The overall aim of the study is to assess the effect of Cerebrolysin on physical and mental development of preterm infants by Denver Scale II at different ages of 5, 7 and 12 months

DETAILED DESCRIPTION:
There is an inverse relationship between birth weight or gestational age and risk for developmental impairment, with increasing incidence as birth weight or gestational age decreases.

Serious impairment, defined as problems in body function or structure which may be temporary or permanent, is generally a more stable condition and typically leads to a disability requiring rehabilitation. Mild impairment is a more reversible condition amenable to early intervention. Studies that have followed extremely preterm and extremely low birth weight infants into school age and early adulthood have shown higher rates of motor, cognitive or behavioral impairments as compared with infants born at term. The neurologic consequences of extreme prematurity range from mild behavioral and cognitive defects to severe disability. Perinatal neuroprotection aims to reduce these outcomes.

Cerebrolysin is a porcine brain-derived peptide preparation that acts like endogenous neurotrophic factors. It is produced by a standardized enzymatic breakdown of lipid-free brain protein powder and consists of low molecular weight peptides and free amino acids.

The pharmacodynamic effects of Cerebrolysin can be categorized in terms of neuronal survival (e.g. trophic and survival promoting actions), neuroprotection (e.g. limiting neuronal dysfunction, especially in adverse conditions), neuroplasticity (e.g. adaptive responses to changing conditions) and neurogenesis (e.g. promoting differentiation of progenitor cells). We aim to assess the effect of Cerebrolysin on physical and mental development of preterm infants at different ages of life at 5, 7 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* High risk preterm infants born with gestational age less than 32 weeks and have a corrected postnatal age of 5 months at time of enrollment. Included preterm infants should have one or more of the following risk factors which may affect their neurodevelopmental outcome.

  1. Infants diagnosed with bronchopulmonary dysplasia requiring oxygen therapy more than 30% FIO2 at 36 weeks corrected gestational age.
  2. Infants with culture proven early or late onset neonatal sepsis with or without neonatal meningitis.
  3. Infants diagnosed to have peri- ventricular leukomalacia diagnosed by brain imaging.

Exclusion Criteria:

1. Patient with persistent uncontrolled fits (all possible reasons for these uncontrolled seizures, including non-epileptic seizures, pseudo intractability, and medically refractory epilepsy.
2. Patient with brain malformation.

Ages: 5 Months to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Neurodevelopmental outcome | 9 months
  Assessment of the physical and mental functions of preterm infant by Denver Developmental Screening Test II (DDST II)

SECONDARY OUTCOMES:
Side effects of cerebrolysin therapy | 9 months
  Sweating, dizziness, increased heart rate and arrhythmia, loss of appetite, diarrhea, constipation, nausea, irritability, insomnia, and allergic reactions.

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University Children Hospital, Al Mansurah, El Dakahlya, Egypt

IPD SHARING:
Plan to Share IPD: Undecided